CLINICAL TRIAL: NCT03161470
Title: Efficacy of a Mechanical Chair for Treatment of Benign Paroxysmal Positional Vertigo (BPPV)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Physicians/audiologists preferred to manage patients with BPPV immediately rather than enrolling in study except for difficult to treat cases.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Richard A. Roberts, Ph.D., Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160176
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Vertigo; Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Vertigo; Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Repositioning (Active Comparator): Participants randomly selected for this treatment arm will undergo standard BPPV treatments (canalith repositioning procedure) without the mechanical chair.
  Interventions: Other: Standard Repositioning
- Mechanical Chair Repositioning (Experimental): Participants randomly selected for this treatment arm will undergo standard BPPV treatments (canalith repositioning procedure) with the mechanical chair.
  Interventions: Other: Mechanical Chair Repositioning
- Sham Treatment (Sham Comparator): Participants randomly selected for the sham arm will undergo be strapped into the mechanical chair as for the treatment arm but will only undergo the test positions for BPPV-the Dix-Hallpike maneuver. No BPPV repositioning treatment will be completed at the first encounter. At the follow-up visit, standard BPPV treatments (canalith repositioning procedure) will be completed.
  Interventions: Other: Sham Treatment

INTERVENTIONS:
Other: Standard Repositioning — It is standard clinical practice for patients with BPPV to undergo treatment by moving the patient through specific head/body positions which moves the displaced otoconial debris out of the involved area of the inner ear.
  Other Names: Epley Maneuver; Semont Liberatory Maneuver; BPPV Treatment Maneuver
  Arms: Standard Repositioning
Other: Mechanical Chair Repositioning — It is standard clinical practice for patients with BPPV to undergo treatment by moving the patient through specific head/body positions which moves the displaced otoconial debris out of the involved area of the inner ear.
  Other Names: Epley Maneuver; Semont Liberatory Maneuver; BPPV Treatment Maneuver
  Arms: Mechanical Chair Repositioning
Other: Sham Treatment — Participants will be placed into the mechanical chair and moved into various positions that do not treat BPPV.
  Arms: Sham Treatment

SUMMARY:
Benign paroxysmal positional vertigo (BPPV) is the most common inner ear cause of dizziness. It has been reported that up to 900 of every 10,000 people in the United States experience this problem with an estimated annual healthcare cost approaching $2 Billion. This problem occurs when calcium carbonate "crystals" which are present and needed in one part of the balance area of the inner ear become displaced to a different part of the balance area. This is very disruptive to the function of the inner ear and results primarily in intense vertigo. Nausea,imbalance, and falls can also occur. The accepted course of management for BPPV is the use of "repositioning maneuvers" which are completed by moving patients through specific head/body positions that literally reposition the displaced crystals out of the wrong area. These treatment methods are reported to be effective for about 80% of patients after one-to-three treatments. For the remaining 20% of patients, more treatments may be necessary and for a small percentage of patients surgical options may be the only cure. Additionally, some patients with BPPV are not able to physically move into the needed positions because of hip and neck problems, spinal problems, obesity, other mobility limitations, etc. Within the past decade, a motorized chair was developed to help reposition any patient with BPPV. There have been no reported adverse incidents with the motorized chair but the device was quite expensive so it was only available at a handful of clinical sites. At this time the motorized chair is no longer being manufactured. More recently, a mechanical chair was developed and has been in use in Europe and China. The mechanical chair has all the advantages of the motorized chair but with a lesser cost. The inventor of the mechanical chair has also developed some slight variations on treatment technique that may have the potential to improve treatment efficacy. We are privileged to have the only mechanical chair of this type in the United States. The primary purpose of the current project is to systematically investigate the treatment efficacy of this mechanical chair for patients with BPPV. We will compare treatment outcomes for patients diagnosed with BPPV using standard methods, the mechanical chair, and a sham condition also using the mechanical chair. A secondary purpose is to determine treatment efficacy for patients with covert BPPV. We will simply measure if treatment with the mechanical chair has any effect on patient symptoms. If we determine treatment is improved with the mechanical chair then it may be possible to help a greater number of patients with BPPV with fewer treatments.

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo (BPPV) is the most common cause of vertigo (Bhattacharyya et al., 2017). BPPV is estimated to affect 900 out of 10,000 people annually (Kerrigan et al., 2013) with healthcare costs approaching $2 Billion (Bhattacharyya et al., 2017). We have shown that patients with BPPV rate the impact on their quality of life similar to patients with macular degeneration, hepatitis B, and HIV/AIDS (Roberts et al., 2009). BPPV occurs when calcium carbonate crystals from one part of the inner ear balance system (utricle) become displaced into other parts of the inner ear balance system (semicircular canal). Normal head and body movements cause movement of the crystal debris within the semicircular canals. This movement causes changes in stimulation of the sensory structures of the semicircular canals that result in vertigo, nausea, imbalance, and even falls. It is well established that BPPV affects the posterior semicircular canal 80% of the time, the horizontal canal 15% of the time and the anterior canal 5% of the time.

There are established methods that have been proven to be effective in treatment of BPPV with randomized controlled trials (Hilton & Pinder, 2014). Each of these methods involves moving a patient's head and body through specific positions to remove the debris from the involved canal. However, many of these patients require multiple treatments and there is a group of patients with BPPV that do not respond to these treatments and for whom surgical options are ultimately considered. Further, patients with hip or neck problems, spinal issues, and even obesity are often unable to be placed in or move through the required positions.

A motorized chair was developed to improve treatment consistency and efficacy and broaden the group of patients who could receive appropriate treatment (Nakayama & Epley, 2005). Although the motorized chair was effective and there are no known reports of adverse events, it was also very expensive. Few facilities were able to purchase the motorized chair so the anticipated impact on helping patients with BPPV was never realized. The motorized chair is no longer being manufactured. A mechanical chair for assessment and treatment of BPPV was also described around the same time as the motorized chair (Richard-Vitton et al., 2005). This is referred to as the TRV chair which are the initials of the inventor.

This mechanical chair has been used in several countries including across Europe and in China. Wang et al. (2014) reported they were able to clear various types of BPPV in 202 of 208 (97.1%) cases. The remaining six cases reported significant improvement. There was no control group in this study and the inventor is listed as an author. No adverse events were reported. West et al. (2016) completed a retrospective chart review of patients treated for BPPV in their clinic.Interestingly, they had both the TRV chair and the motorized chair. Some of their patients also underwent treatment with traditional methods which do not incorporate a specialized chair to help position patients. The authors concluded that specialized chairs (motorized or mechanical) are useful for treatment of BPPV, especially for more difficult cases. There are also some limitations with this report in that no control group was used and participants were not randomly assigned to a treatment type. Patients with a typical history of BPPV, and identified with the most common type affecting the posterior canal, were treated with the traditional methods first and then perhaps with a specialized chair. Other patients were treated with both types of chair. No adverse events were reported.

Specialized chairs do appear to offer some advantages over traditional methods of BPPV treatment. Reports in the literature suggest the specialized chairs are able to treat more difficult cases of BPPV. This should allow improved cure rates for the approximately 20% of patients that require multiple treatments using the traditional methods. Use of specialized chairs would also increase the number of patients who can be treated because there are no contraindications related to hip, spine, and mobility issues as there are for traditional methods of BPPV treatment. The mechanical chair (TRV chair) appears to offer all of the advantages of the motorized chair but at a lessor cost anticipated to be $65,000 compared to $100,000 for the motorized chair. One may speculate there is less maintenance required for a mechanical versus a motorized system and there is the fact that the currently described motorized version is no longer available for purchase.

The primary purpose of this project is to determine treatment efficacy of the motorized TRV chair for patients with BPPV. This information has not been published using a randomized controlled design. A secondary purpose of the project is to determine if the TRV chair is helpful in patients experiencing chronic symptoms of dizziness and unsteadiness who may have complaints suggesting positional vertigo but who fail to generate nystagmus (i.e. covert BPPV). If the TRV chair is more efficacious than traditional methods, our hope is that nearly all patients with BPPV will be able to be managed in a more efficient manner. This will decrease the impact of BPPV on health-related quality of life, could decrease falls related to BPPV, and should also decrease the burden of healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients identified with BPPV through the Vanderbilt Balance Disorders Clinic or diagnosed with BPPV by Vanderbilt Otolaryngology will be eligible for inclusion.

Exclusion Criteria:

* Patients without BPPV. Also, the mechanical chair is contraindicated for for patients weighing over 330 lbs, patients presenting with unusual headache symptoms, uncontrolled high blood pressure or some associated neurological symptoms or any other atypical findings. It must not be used if the patient has undergone neurosurgery or cardiac surgery within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Dix-Hallpike Test | Treatment will take 15 minutes. Patient will be assessed seven days later.
  This is the test used to determine if a patient is positive or negative for posterior or anterior canal BPPV.
Roll Test | Treatment will take 15 minutes. Patient will be assessed seven days later.
  This is the test used to determine if a patient is positive or negative for horizontal canal BPPV.

SECONDARY OUTCOMES:
Dizziness Handicap Inventory | Ten minutes before intervention and seven days after intervention.
  This is a validated subjective measure of impact of dizziness on health-related quality of life.
Percent Dizziness is Improved | Five minutes before treatment and seven days post-treatment
  Patients will rate their dizziness on a zero to 100 point scale. Zero will be no dizziness and 100 will be maximum dizziness.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No